CLINICAL TRIAL: NCT04950140
Title: Randomized Clinical Trial Comparing Conventional Laparoscopic Surgery and Robot-Assisted Laparoscopic Surgery for the Treatment of Parastomal Hernia of the Oncology Patient
Acronym: LAROPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP1465
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Parastomal Hernia; Oncology
MeSH Terms: conditions — Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Robot Assisted Laparoscopic (Experimental): Robot Assisted Laparoscopic Surgery for the Treatment of Parastomal Hernia of the Oncology Patient
  Interventions: Procedure: Robot Assisted Laparoscopic Surgery for the Treatment of Parastomal Hernia
- Conventional Laparoscopic Surgery (Active Comparator): Conventional Laparoscopic Surgery for the Treatment of Parastomal Hernia of the Oncology Patient
  Interventions: Procedure: Laparoscopic Surgery for the Treatment of Parastomal Hernia

INTERVENTIONS:
Procedure: Robot Assisted Laparoscopic Surgery for the Treatment of Parastomal Hernia — Robot Assisted Laparoscopic Surgery for the Treatment of Parastomal Hernia of the Oncology Patient
  Arms: Robot Assisted Laparoscopic
Procedure: Laparoscopic Surgery for the Treatment of Parastomal Hernia — Laparoscopic Surgery for the Treatment of Parastomal Hernia in Cancer Patients
  Arms: Conventional Laparoscopic Surgery

SUMMARY:
Prospective randomized prospective interventional study with 40 consecutive patients for whom surgical treatment for PH was indicated and who are in postoperative follow-up with the Oncology Surgery group of the Department of Digestive Tract Surgery and Coloproctology, Faculty of Medicine, University of São Paulo .

The free and informed consent form will be applied to the patient by the researchers in two copies of equal content and after any doubts related to the research are resolved, the patient will sign the copies together with the researcher. At any time, the patient may opt out of the study. The contacts of the researchers and the institution will be fully available to the research subject to resolve doubts and for any eventuality that may occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PH in permanent ostomy, aged between 18 and 75 years, undergoing surgery for cancer treatment at ICESP, with stable cancer disease (recurrence or metastasis without evolution) or in follow-up after treatment with curative intent, who have computed tomography with a diagnosis of HP, and who agree to participate in the study.

Exclusion Criteria:

* Patient with progressive cancer disease. Presence of disease that prevents the performance of videolaparoscopic surgical procedure such as severe heart failure, severe lung disease, etc. Clinical criteria according to the research team that may indicate the application of another specific technique that is not covered in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-24 (Estimated); Primary Completion 2021-09-24 (Estimated); Study Completion 2023-07-24 (Estimated)

PRIMARY OUTCOMES:
To study the return time of ostomy functioning of patients approached by laparoscopic assisted robot using the Sugarbaker technique using a semi-absorbable biosynthetic mesh. | 1 year

IPD SHARING:
Plan to Share IPD: Yes